CLINICAL TRIAL: NCT04729062
Title: US Early Access Program for the Treatment of Patients With C3 Glomerulopathy or Primary Immune-Complex Membranoproliferative Glomerulonephritis With Pegcetacoplan
Brief Title: C3G/Primary IC-MPGN EAP
Status: Approved for marketing | Type: Expanded Access
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: APL2-C3G-801
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-07

CONDITIONS: C3G; IC-MPGN; C3 Glomerulopathy; C3 Glomerulonephritis; Complement 3 Glomerulopathy; Complement 3 Glomerulopathy (C3G); Complement 3 Glomerulonephritis; Dense Deposit Disease; DDD; Membranoproliferative Glomerulonephritis; Membranoproliferative Glomerulonephritis (MPGN); Immune Complex Membranoproliferative Glomerulonephritis (IC-MPGN)
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — pegcetacoplan

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor

SUMMARY:
This is an Early Access Program (EAP) which will provide access to pegcetacoplan for eligible participants with C3G and Primary IC-MPGN.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged at least 12 years or older weighing at least 30 kg.
2. A biopsy has confirmed diagnosis of primary C3G or IC-MPGN or patient has a biopsy-proven histologic recurrence in posttransplant.
3. There is evidence of active renal disease, based on at least 1 g/day of proteinuria from 24-hour urine collection or uPCR ≥1 g/g from random urine in native kidney. There is no minimum level of proteinuria for post-transplant recurrence.
4. Patient has a limited response to treatment regimens for C3G/IC-MPGN, and may include:

   1. Angiotensin-converting enzyme inhibitor, angiotensin receptor blocker, and/or sodium-glucose cotransporter-2 inhibitor therapy
   2. Other medications that can affect proteinuria (eg, steroids, mycophenolate mofetil, and/or other immunosuppressants that the patient is receiving for treatment of C3G or IC-MPGN)
5. Patient has received vaccinations against S pneumoniae, N meningitidis (types A, C, W, Y, and B), and H influenzae (type B) as per the Advisory Committee on Immunization Practices (ACIP) recommendations for adults or children with complement deficiencies. Vaccination series should be initiated at least 14 days prior to enrollment. If patient disease is severe and requires immediate treatment, administer required vaccine as soon as possible and provide patients with 2 weeks of prophylactic antibiotics.
6. Female patients of childbearing potential, defined as any women who have experienced menarche and who are not permanently sterile or postmenopausal, must have negative blood pregnancy tests at screening (and negative urine pregnancy tests on day 1) and must agree to use protocol-defined methods of contraception from screening through at least 90 days after receiving the last dose of pegcetacoplan.
7. Patients above the legal age of consent, in accordance with local regulations, must be willing and able to provide informed consent. The legally authorized representative of patients under the legal age of consent must be willing and able to provide informed consent; where appropriate, patients under the legal age of consent must also give their assent to participation in the program.
8. Patient is willing and able to self-administer pegcetacoplan or have an identified caregiver who can perform the administration.
9. Patient currently resides in and is a resident of the US.

Exclusion Criteria:

1. C3G/IC-MPGN is secondary to another condition (eg, infection, malignancy, monoclonal gammopathy, a systemic autoimmune disease such as systemic lupus erythematosus, chronic antibody-mediated rejection, or a medication), in the opinion of the treating physician.
2. Patient has current or prior diagnosis of HIV, hepatitis B, or hepatitis C infection or positive serology during screening that is indicative of infection with any of these viruses.
3. Patient's body weight is greater than 100 kg at screening.
4. Patient has hypersensitivity to pegcetacoplan or to any of the excipients.
5. Patient has history of meningococcal disease.
6. Patient has a severe infection (eg, requiring IV antibiotic therapy) within 14 days prior to the first dose of pegcetacoplan.
7. Patient has an absolute neutrophil count less than 1000 cells/mm3 at screening.
8. Patient has other significant renal disease.
9. Based on the investigator's opinion, the patient has significant glomerulosclerosis or interstitial fibrosis on kidney biopsy.
10. Patient is participating in any other investigational drug trial.
11. Patient is a female who is pregnant or who is currently breastfeeding.
12. Patient has the inability to cooperate or has any condition that, in the opinion of the treating physician, creates an undue risk for the patient by participating in the program.
13. There is evidence of ongoing drug or alcohol abuse or dependence, in the opinion of the treating physician.
14. There is the presence or suspicion of severe infection during the screening period (including but not limited to recurrent or chronic infections) that, in the opinion of the treating physician, may place the patient at unacceptable risk by program participation.
15. There is a known or suspected hereditary fructose intolerance.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult